CLINICAL TRIAL: NCT02232061
Title: Long-term, Open-label, Multicenter Study Assessing Long-term Cardiovascular Risks in Patients Treated With Fingolimod
Brief Title: Long-term, Open-label, Multicenter Study Assessing Long-term Cardiovascular Risks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CFTY720D2409
Record Dates: First submitted 2014-09-02; First posted 2014-09-04 (Estimated); Results first posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-01

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis, fingolimod, adult, FTY720, inflammatory disease, demyelination, auto-inflammatory disease, relapsing-remitting MS, CFTY720D2406
MeSH Terms: conditions — Multiple Sclerosis; Demyelinating Diseases | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fingolimod (Experimental): Fingolimod 0.5mg/day tablets taken orally.
  Interventions: Drug: Fingolimod

INTERVENTIONS:
Drug: Fingolimod — Fingolimod 0.5 mg tablet
  Other Names: FTY720

SUMMARY:
This study will evaluate if patients who had a serious cardiovascular event upon initiation of fingolimod are at risk to delevop long term other cardiovascular events

DETAILED DESCRIPTION:
This was a multi-national, long-term safety study. Patients enrolled in study FTY720D2406 who experienced a cardiovascular event within 24-hours of fingolimod treatment initiation which led to overnight monitoring or met serious adverse event criteria, were eligible to participate in this study.

Patients who experienced a qualifying event in study CFTY720D2406 started study CFTY720D2409 approximately 6 months after the occurrence of the CFTY720D2406 qualifying event.

Patients underwent mandatory assessments on a 6-monthly basis including 12-lead ECG, vital signs. Other assessments were performed as per routine practice.

The primary objective of the study was to estimate the long-term cardiovascular risk of fingolimod in patients who experienced a cardiovascular event during treatment initiation.

The study has no stand-alone secondary objective. However data from the CFTY720D2409 and CFTY720D2406 studies will be pooled to supplement CFTY720DD2406 study and support its primary and secondary objectives of evaluating the safety profile of fingolimod.

The pooled data will be appended to this result upon completion of FDA submission.

ELIGIBILITY:
Inclusion Criteria:

* Patients participating in study FTY720D2406 who experienced a serious cardiovascular event during their fingolimod treatment initiation or re-initiation which led to overnight monitoring or met seriousness criteria.
* Patients still on fingolimod after the this first dose serious event

Exclusion Criteria:

-Treatment with any investigational drug unless it is received as part of a Novartis sponsored MS study lasting less than 1 month

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-09-29 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Belgium (2):
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Hasselt
- Novartis Investigative Site, Ravensburg, Germany
- Novartis Investigative Site, Napoli, Italy

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on
  https://www.clinicalstudydatarequest.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients enrolled in study CFTY720D2406 who experienced a cardiovascular event within 24-hours of fingolimod treatment initiation/re-initiation which led to overnight monitoring or met serious adverse event criteria, were eligible to participate in this study CFTY720D2409.
Period: Overall Study
Arm/Group | Fingolimod
Started | 6
Completed | 4
Not Completed | 2
Not completed — Administrative problems | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fingolimod
Number analyzed (Participants) | 6
Age, Customized [Number; unit: participants]
  Ages 21 - 47 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 6

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Experienced at Least One Qualifying Cardiovascular Adverse Event
Description: Participants from study CFTY720D2406 who experienced a qualifying cardiovascular adverse event were transferred to this study. Qualifying cardiovascular events included, but were not limited to, sudden unexplained death, cardiovascular death, myocardial infarction (MI), Q-wave MI, stroke (ischemic or hemorrhagic), unstable angina requiring hospitalization, congestive heart failure requiring hospitalization, complete heart block, ventricular fibrillation, torsade de pointes, hypertensive emergency and any other suspected life threatening cardiovascular condition.
Time Frame: Within 6 months of qualifying event up to 64 months
Measure: Number; unit: participants
Arm/Group | Fingolimod
Number analyzed (Participants) | 6
participants | 0

ADVERSE EVENTS:
Time Frame: Within 6 months of qualifying event up to approximately 64 months
Arm/Group | Fingolimod
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod (N=6)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1
BRONCHITIS VIRAL (Infections and infestations) | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod (N=6)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1
HYPOTHYROIDISM (Endocrine disorders) | 1
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1
PYREXIA (General disorders) | 1
NASOPHARYNGITIS (Infections and infestations) | 1
TRICHOMONIASIS (Infections and infestations) | 1
VIRAL PHARYNGITIS (Infections and infestations) | 1
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1
FOLATE DEFICIENCY (Metabolism and nutrition disorders) | 1
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 1
HYPERPHAGIA (Metabolism and nutrition disorders) | 1
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1
BURSITIS (Musculoskeletal and connective tissue disorders) | 1
FACET JOINT SYNDROME (Musculoskeletal and connective tissue disorders) | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1
HEADACHE (Nervous system disorders) | 1
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 1
SCIATICA (Nervous system disorders) | 1
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1
ANXIETY (Psychiatric disorders) | 1
INSOMNIA (Psychiatric disorders) | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1
HOT FLUSH (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
This study had no stand-alone secondary objectives. However, data from the CFTY720D2409 and D2406 studies will be pooled to supplement this study and will be appended to this record when available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT02232061/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT02232061/SAP_001.pdf